CLINICAL TRIAL: NCT02787824
Title: Periodic Versus Continuous (at Every Session of Hemodialysis) iv Iron Supplementation in Chronic HD Patients
Brief Title: Periodic Versus Continuous IV Iron Supplementation in HD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Papageorgiou General Hospital (Other)
Responsible Party: Principal Investigator, Efstathios Mitsopoulos, Director of Nephrology Dept, Papageorgiou General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 637/13.7
Record Dates: First submitted 2016-05-24; First posted 2016-06-01 (Estimated); Last update posted 2017-09-20 (Actual); Status verified 2016-05

CONDITIONS: Anemia of Chronic Kidney Disease
Keywords: iron deficiency; hemodialysis
MeSH Terms: conditions — Iron Deficiencies

ARMS (2):
- continuous iv administration of iron sucrose (Experimental): Prior to the study, all our patients were receiving intravenous iron sucrose in an intermittent mode (every 1-4 weeks).Patients on this arm will receive the same previous dose of iron glucose but in a continuous mode (smaller doses of iron sucrose in every session).
  Interventions: Drug: Iron Sucrose Supplement
- intermittent iv administration of iron sucrose (Active Comparator): Patients on this arm will continue to receive the same previous intermittent mode of iron sucrose.
  Interventions: Drug: Iron Sucrose Supplement

INTERVENTIONS:
Drug: Iron Sucrose Supplement

SUMMARY:
The purpose of this study was to compare the efficacy of two regimens of intravenous iron sucrose [continuous (in every hemodialysis session) versus intermittent (every 1-4 weeks)] on the response of rHuEPO in the maintenance phase of its administration in hemodialysis patients.

ELIGIBILITY:
Inclusion Criteria:

* Constant rHu-EPO and iron dose for at least 2 months before starting the study
* Hemoglobin ≥ 8,5g/dl and <12,5 g/dl
* Ferritin < 1000 mg/dl
* TSAT < 50%
* CRP < 5 mg/dl

Exclusion Criteria:

* Malignant tumor disease
* Oral iron supplementation
* Active bleeding issues
* Surgical intervention within the last 8 weeks before study inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-05; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change of serum hemoglobin level (g/dl) | Month 0, 1, 2, 3, 4

CONTACTS AND LOCATIONS:
Locations (1):
- Papageorgiou General Hospital, Thessaloniki, Greece